CLINICAL TRIAL: NCT03785275
Title: Beta Cell Imaging in Type 1 Diabetes With Stable Near-normal and Unstable Glucose Control Using PET
Brief Title: Beta Cell Imaging in T1D Patients With a Different Glycemic Control
Acronym: GLP1-reg
Status: Terminated | Type: Observational
Why Stopped: It was not possible to include 9 study participants with unstable glucose in due time, and therefore 7 individuals with unstable glucose control were included.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL59582.091.17
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with stable near-normal T1D: * Mixed-meal tolerance test
  * Intravenous injection with gallium-68-exendin followed by a PET/CT scan
  Interventions: Radiation: gallium-68-exendin PET/CT
- Subjects with unstable T1D: * Mixed-meal tolerance test
  * Intravenous injection with gallium-68-exendin followed by a PET/CT scan
  Interventions: Radiation: gallium-68-exendin PET/CT

INTERVENTIONS:
Radiation: gallium-68-exendin PET/CT — PET/CT scan after injection with gallium-68-exendin

SUMMARY:
The primary aim of this study is to measure (residual) beta cell mass in type 1 diabetes (T1D) patients with stable near-normal and unstable glucose control using PET/CT imaging, to improve the understanding of the relation between beta cell mass and glycemic control in T1D.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is characterized by a progressive decrease in beta cell function due to an autoimmune attack on the beta cells, which will lead to a reduction in insulin secretion. Endogenous insulin secretion can be determined measuring C-peptide, which is secreted in equal amounts to insulin. The loss of insulin secretion, indicated by an immeasurable C-peptide level, will hamper glycemic control which results in increased glycated haemoglobin (HbA1c) levels. Also, hypoglycemic events can occur more frequently. Initially, the belief was that this could be explained by the loss of all pancreatic beta cells due to the autoimmune attack. However, recent literature suggests that a considerable number of beta cells can survive this attack. This could mean that certain beta cells survived, but have lost their function. The ratio of functional and non-functional residual beta cells might play an important role in the degree of glycemic control. It would therefore be of great interest to study residual beta cell mass in two types of T1D patients that differ in glycemic control. Although both types of patients receive treatment, one group of patients is characterized by a stable near-normal glucose control while the second group is characterized by an unstable glucose control. In case glycemic control mostly depends on beta cell function and less on beta cell mass, novel therapies could focus on the functional reactivation of these non-functional beta cells to restore overall beta cell function. This could especially be in favour of patients with an unstable glucose control. Beta cell mass will be determined using Ga-68-NODAGA-exendin-4 positron emission tomography (PET), which allows visualization of pancreatic beta cells as well as absolute quantification of tracer uptake, providing a measure for the pancreatic beta cell mass. The outcome of this study will lead to a better understanding of the relation between the amount of residual beta cells, beta cell function and the influence of glycemic control. This could provide new insights regarding the development of new therapies to improve beta cell function and glycemic control, which could lower disease burden and improve the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (stable glycemic control)

* Age ≥18 years
* T1D diagnosed ≥1 year at the start of the study
* HbA1c <7 (<53 mmol/mol)
* 17≤ BMI ≤30 kg/m2
* No severe hypoglycemic events in the past year and a maximum of 2 severe hypoglycemic events in their entire life.
* Intact hypoglycemic awareness
* Ability to sign informed consent

Group 2 (unstable glycemic control) Age ≥18 years

* T1D diagnosed ≥1 year at the start of the study
* HbA1c >8.5 (>69 mmol/mol)
* 17≤ BMI ≤30 kg/m2
* Minimum of 2 severe hypoglycemic events in the past year, or an impaired awareness of hypoglycemia (subjects may comply with both criteria, but this is not a requirement)
* Ability to sign informed consent

Exclusion Criteria:

* Previous treatment (within 6 months) with synthetic Exendin (Exenatide, Byetta®) or Dipeptidyl-Peptidase IV inhibitors
* Liver disease
* Renal disease
* Pregnancy or the wish to become pregnant within 6 months after the study
* Breastfeeding
* BMI <17 kg/m2 or BMI >30 kg/m2
* Age <18 years
* Inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include 18 individuals with T1D for at least 1 year with a minimum age of 18 years. This population consists of two groups that include 9 subjects with stable near-normal glucose control and 9 individuals with unstable glucose control. The differentiation between T1D patients with stable near-normal and unstable glucose control will be based on their HbA1c value, the number of severe hypoglycemic events and the patient's hypoglycaemic awareness.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Beta cell mass | 2 years
  Pancreatic uptake of the tracer is measured by quantitative analysis (measure for beta cell mass)

SECONDARY OUTCOMES:
Beta cell mass vs. beta cell function | 2 years
  The correlation of the measured beta cell mass to the beta cell function

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands